CLINICAL TRIAL: NCT04309890
Title: Validating 7-items Overactive Bladder Symptom Score (OABSS) Through Arabic Linguistic Version
Brief Title: Arabic Translation and Validation of the (Overactive Bladder Symptom Score) OABSS
Status: Completed | Type: Observational
Sponsor: Mutah University (Other)
Responsible Party: Principal Investigator, Fadi Sawaqed, Dr, Mutah University
Other Study IDs: Arabic OABSS- 7 items
Record Dates: First submitted 2020-03-13; First posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group
  Interventions: Other: Arabic version of the Overactive Bladder Symptom Score Questionnaire

INTERVENTIONS:
Other: Arabic version of the Overactive Bladder Symptom Score Questionnaire — All enrolled patients were asked to complete the Arabic OABSS questionnaire in its final edition before and three months after treatment with Solfinasin 5 mg once daily

SUMMARY:
The English version of the Overactive Bladder Symptom Score (OABSS) questionnaire was translated to Arabic language. The questionnaire was validated by comparing the response to the questionnaire in a patient with Overactive Bladder (OAB) before and after providing treatment with antimuscarinics.

ELIGIBILITY:
Inclusion Criteria:

* More than 20 years
* Had three months history of overactive bladder symptoms (urgency with or without incontinence and associated with frequency and nocturia).

Exclusion Criteria:

* Active urinary tract infection.
* Predominant symptoms of urinary stress incontinence;
* Diabetes mellitus;
* Previous abdominal and pelvic (urological or gynecological gastrointestinal) surgery;
* Previous neurological disease.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study has included 235 patients, 152 (62.9%) females and 83 (37.1%) males.
Sampling Method: Non-Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
development and validation of Arabic version of the Overactive Bladder Symptom Score (OABSS) questionnaire | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Mu'tah University, Karak, Jordan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sawaqed F, Suoub M. Validating 7-items Overactive Bladder Symptom Score (OABSS) through Arabic linguistic version. Sci Rep. 2021 Jan 12;11(1):661. doi: 10.1038/s41598-020-79974-9. PMID 33436744